CLINICAL TRIAL: NCT03311451
Title: Clinical Trial To Evaluate Safety and Dose Response Using the C2 CyroBalloon™ 180 Ablation System for the Treatment of Dysplastic Barrett's Esophagus.
Brief Title: C2 CryoBalloon™ 180 Ablation System Dose De-escalation Study.
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Pentax Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP-0019
Record Dates: First submitted 2017-10-10; First posted 2017-10-17 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Barrett Esophagus
MeSH Terms: conditions — Barrett Esophagus

STUDY DESIGN:
Intervention Model Description: Patients with previously untreated (by means of ablation therapy) flat type Barrett's Esophagus (BE) (extent BE ≤C3 and ≥M1) with Low-Grade Dysplasia (LGD) or High-Grade Dysplasia (HGD), or residual BE after endoscopic resection of dysplasia or early adenocarcinoma.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- C2 CryoBalloon 180 Ablation System (Other): C2 CryoBalloon 180 Ablation System will be used to ablate visible Barrett's esophagus
  Interventions: Device: C2 CryoBalloon 180° Ablation System

INTERVENTIONS:
Device: C2 CryoBalloon 180° Ablation System — The C2 CryoBalloon 180° Ablation System is a cryosurgical device with a nitrous oxide cooled balloon probe that is compatible with upper gastrointestinal therapeutic endoscopes.
  Other Names: CryoBalloon 180

SUMMARY:
The primary objective is to determine the safety, performance and efficacy of the C2 CryoBalloon 180 Ablation System ("CryoBalloon 180") used at decreasing doses in treatment naïve patients with low- or high-grade dysplastic Barrett's Esophagus (BE) or with residual BE after resection of dysplasia or early adenocarcinoma.

DETAILED DESCRIPTION:
The procedure will be performed on an outpatient basis, and the CryoBalloon 180 Ablation system will be used for all ablations following the instructions for use provided with the product.

Patients who meet the eligibility criteria will be assigned to one of the treatment groups and doses, depending on the order of their enrollment:

In phase I, the first 25 patients will be treated with Dose 1 (lowest), in one application to ablate 50% of the esophageal circumference.

All patients will undergo 10 week (±2 weeks) follow-up EGD to evaluate efficacy of the dose before the study continues.

If follow-up shows that Dose 1 eradicates ≤60% of the treated BE (by median percentage) and no SAE's are reported, the treatment phase will continue but at the next incremental higer dose (Second Dose) after approval from the IRB.

If the Dose 1 median BE surface regression percentage is ≥60%, the dose is defined as the therapeutic dose. In that case, an additional group of 25 patients will be enrolled at this dose, pending IRB approval.

---------------------------------------------------------------

Dose-related SAEs include pain in the treatment area greater than 6 (0-10 VAS score) at 24 hours AND seven (7) days post-treatment; symptomatic stricture requiring an additional EGD with endoscopic dilation before the first follow-up EGD; symptomatic stricture at follow-up EGD; or any stricture (symptomatic or asymptomatic) preventing passage of the therapeutic endoscope at follow-up EGD. Any other serious adverse events within 30 days after treatment will also be evaluated by the Data and Safety Monitoring Board (DSMB) for relationship to the dose and severity.

When a Dose-related serious adverse event occurs, the Holding Rule will be invoked and enrollment at that dose will be held until the DSMB has evaluated the event.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with flat- type BE esophagus, with an indication for ablation therapy, defined as:

   * Diagnosis of LGD or HGD in BE (confirmed by central pathology review), OR
   * Residual BE with any grade of dysplasia 6 weeks after endoscopic resection
2. Prague Classification Score C≤3 and ≥M1
3. Patients should be ablation-naïve (no previous ablation therapy of the esophagus)
4. Older than 18 years of age at time of consent
5. Operable per institution's standards
6. Patient provides written informed consent on the IRB-approved informed consent form
7. Patient is willing and able to comply with follow-up requirements.

Exclusion Criteria:

1. Esophageal stenosis preventing advancement of a therapeutic endoscope
2. Any endoscopically visualized lesion such as ulcers, masses or nodules. Neoplastic nodules must first be treated with ER >6 weeks prior to planned treatment under this protocol.
3. Prior ER of more than 2cm in length or >50% of the esophageal lumen circumference
4. History of locally advanced (>SM1) esophageal cancer
5. History of esophageal varices
6. Prior distal esophagectomy
7. Active esophagitis LA grade B or higher
8. Severe medical comorbidities precluding endoscopy
9. Uncontrolled coagulopathy
10. Pregnant or planning to become pregnant during period of study
11. Patient refuses or is unable to provide written informed consent
12. Participation in another study with investigational drug within the 30 days preceding or during the present study, interfering with participation in the current study
13. General poor health, multiple co-morbidities placing the patient at risk or otherwise unsuitable for trial participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-01-16 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Efficacy: Dose response | 10 weeks
  Dose response (efficacy) is defined as eradication percentage of BE confirmed by histological evidence of eradication of BE, after treatment with the therapeutic dose (phase II).
Safety: Incidence of Dose-related SAEs | 30 days
  Safety will be evaluated by the incidence of Dose-related SAEs.
  Dose-related SAEs include pain in the treatment area, or any stricture (symptomatic or asymptomatic) preventing passage of the diagnostic endoscope at follow-up EGD.

SECONDARY OUTCOMES:
Incidence of AEs | 30 days
  Incidence of all serious and non-serious adverse events up to 30 days post-treatment
Patient reported post-procedure pain | 24hours and 7 days post-procedure
  Post-procedure pain in the area of the cryoablation treatment (0-10 VAS score)
Efficacy: Percent Regression | 10 weeks
  Efficacy, defined as the regression percentage at the first follow-up endoscopy, after one (1) treatment covering 50% of circumference of the esophagus with the therapeutic dose.
Efficacy: Treatment | 10 weeks
  Efficacy of treatment with CryoBalloon 180 Ablation system, defined as the proportion of patients with ≥80% regression of BE after 1 hemi-circumferential and after full circumferential treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Bas LA Weusten, MD, PhD, Principal Investigator — St. Antonius Ziekenhuis, Niewegein The Netherlands
Locations (5):
- Netherlands (5):
  - AMC Medical Research B.V., Amsterdam
  - UMC Groningen, Groningen
  - St. Antonius Hospital, Nieuwegein
  - Erasmus Medical Center, Rotterdam
  - UMC Utrecht, Utrecht

IPD SHARING:
Plan to Share IPD: No
Data will not be shared.